CLINICAL TRIAL: NCT04794725
Title: Monitoring Of Viral Load In Decentralised Area 1 Ter - Evaluation of the Cobas® Plasma Separation Card in the Field in Vietnam
Brief Title: MOVIDA 1 Ter - Evaluation of the Cobas® Plasma Separation Card in the Field in Vietnam
Acronym: MOVIDA1-Ter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-067
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: HIV Infections
Keywords: Viral Load Monitoring, Dried Blood Spot
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Sampling (Other): blood samples from venepuncture (10mL)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — blood samples from venepuncture (10mL)

SUMMARY:
In low- and middle-income countries, viral load (VL) monitoring of patients living with HIV and followed on antiretroviral therapy (ART) in remote settings is still scarce. Barriers to VL monitoring are essentially the limited access to a laboratory able to perform this measurement, its cost, as well as the lack of human and material resources. Blood sampling using dried blood spots (DBS), which has been validated and is immediately available, could overcome these barriers. With DBS, transfer and conservation of samples are simplified enabling access to VL monitoring to patients seeking care in sites far from laboratory facilities. Use of DBS also offers the advantage not to require extensive investments.

To guide decision makers in the implementation of strategies to scale-up HIV VL monitoring in remote settings, field evaluations of DBS in routine conditions are needed. It is in this context that we propose this field evaluation of the Cobas® plasma separation card in Vietnam

DETAILED DESCRIPTION:
In Vietnam, in 2018, HIV prevalence was estimated at 0.3% among adults and the estimated proportion of PLHIV on ART was 65%, however the HIV epidemic is essentially concentrated in people who inject drugs, men who have sex with men and sex workers.

As of today, routine HIV VL monitoring is not yet available in remote settings in Vietnam. Despite an initiative we conducted and that documented the feasibility of DBS use in remote settings, and although no genuine roll-out of POC machines is yet observed in the field, the Ministry of Health of Vietnam has not yet decided to scale-up HIV VL monitoring using DBS. More field evaluations are needed to convince the Ministry of Health that DBS can effectively be used to scale-up HIV VL monitoring.

The aim of the present study is to evaluate the sensitivity and specificity of HIV VL measurement using the cobas® plasma separation card (PSC) against plasma at the threshold of 1000 copies/mL (threshold currently used to define failure in Vietnam, following the WHO guidelines).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* HIV-1 infected adults
* Willing to participate to the study by giving his/her consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Quantification of HIV RNA on DBS compared to plasma as gold standard | up to 4 weeks
  sensitivity and specificity of the Cobas® PSC against plasma (as gold standard) at to identify virological failure (HIV VL ≥1000 copies/mL)

SECONDARY OUTCOMES:
Correlation between HIV RNA VL measured on DBS and on plasma | up to 4 weeks
  Comparison of quantitative HIV VL results obtained on plasma and when using the cobas® PSC

CONTACTS AND LOCATIONS:
Overall Officials: Yoann MADEC, PhD, Study Director — Institut Pasteur; Tuan Anh NGUYEN, MD, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (2):
- Vietnam (2):
  - Dong Da, Hanoi
  - Nam Tu Liem, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen TA, Tran TH, Nguyen BT, Pham TTP, Hong Le NT, Ta DV, Phan HTT, Nguyen LH, Ait-Ahmed M, Ho HT, Taieb F, Madec Y; MOVIDA 2 study group. Feasibility of dried blood spots for HIV viral load monitoring in decentralized area in North Vietnam in a test-and-treat era, the MOVIDA project. PLoS One. 2020 Apr 9;15(4):e0230968. doi: 10.1371/journal.pone.0230968. eCollection 2020. PMID 32271796
- [Background] Taieb F, Tran Hong T, Ho HT, Nguyen Thanh B, Pham Phuong T, Viet Ta D, Le Thi Hong N, Ba Pham H, Nguyen LTH, Nguyen HT, Nguyen TT, Tuaillon E, Delaporte E, Le Thi H, Tran Thi Bich H, Nguyen TA, Madec Y. First field evaluation of the optimized CE marked Abbott protocol for HIV RNA testing on dried blood spot in a routine clinical setting in Vietnam. PLoS One. 2018 Feb 9;13(2):e0191920. doi: 10.1371/journal.pone.0191920. eCollection 2018. PMID 29425216